CLINICAL TRIAL: NCT04836195
Title: Phase I Trial of PCLX-001 in Relapsed/Refractory B-cell Non-Hodgkin Lymphoma and Advanced Solid Malignancies
Brief Title: Study of PCLX-001 in R/R Advanced Solid Malignancies and B-cell Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pacylex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PCLX-001-01
Record Dates: First submitted 2021-03-29; First posted 2021-04-08 (Actual); Results first posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: B-cell Non Hodgkin Lymphoma; Advanced Solid Tumor
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: For Part A dose-escalation, patients will be enrolled in cohorts of 3 to 6 patients to each dose level. Six patients will be treated at the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- PCLX-001 intervention 20mg (Experimental): Cohort 1: Participants were administered 20mg of PCLX-001 orally as continuous daily dosing on a 28-day cycle.
  Interventions: Drug: PCLX-001 - 20mg
- PCLX-001 intervention 40mg (Experimental): Cohort 2: Participants were administered 40mg of PCLX-001 orally as continuous daily dosing on a 28-day cycle.
  Interventions: Drug: PCLX-001 - 40mg
- PCLX-001 intervention 70mg (Experimental): Cohort 3: Participants were administered 70mg of PCLX-001 orally as continuous daily dosing on a 28-day cycle.
  Interventions: Drug: PCLX-001 - 70mg
- PCLX-001 intervention 100mg (Experimental): Cohort 4: Participants were administered 100mg of PCLX-001 orally as continuous daily dosing on a 28-day cycle.
  Interventions: Drug: PCLX-001 - 100mg
- PCLX-001 intervention 140mg (Experimental): Cohort 5: Participants were administered 140mg of PCLX-001 orally as continuous daily dosing on a 28-day cycle.
  Interventions: Drug: PCLX-001 - 140mg
- PCLX-001 intervention 210mg (Experimental): Cohort 6: Participants were administered 210mg of PCLX-001 orally as continuous daily dosing on a 28-day cycle.
  Interventions: Drug: PCLX-001 - 210mg
- PCLX-001 intervention 280mg (Experimental): Cohort 7: Participants were administered 280mg of PCLX-001 orally as continuous daily dosing on a 28-day cycle.
  Interventions: Drug: PCLX-001 - 280mg

INTERVENTIONS:
Drug: PCLX-001 - 20mg — 20mg daily oral pills
  Other Names: zelenirstat
  Arms: PCLX-001 intervention 20mg
Drug: PCLX-001 - 40mg — 40mg daily oral pills
  Other Names: zelenirstat
  Arms: PCLX-001 intervention 40mg
Drug: PCLX-001 - 70mg — 70mg daily oral pills
  Other Names: zelenirstat
  Arms: PCLX-001 intervention 70mg
Drug: PCLX-001 - 100mg — 100mg daily oral pills
  Other Names: zelenirstat
  Arms: PCLX-001 intervention 100mg
Drug: PCLX-001 - 140mg — 140mg daily oral pills
  Other Names: zelenirstat
  Arms: PCLX-001 intervention 140mg
Drug: PCLX-001 - 210mg — 210mg daily oral pills
  Other Names: zelenirstat
  Arms: PCLX-001 intervention 210mg
Drug: PCLX-001 - 280mg — 280mg daily oral pills
  Other Names: zelenirstat
  Arms: PCLX-001 intervention 280mg

SUMMARY:
This is a phase I dose-escalation study of oral PCLX-001, conducted in a multicenter, non-randomized, open-label, non-controlled design. The study is comprised of two parts: Part A (single-agent dose escalation) and Part B (single-agent expansion cohorts).

DETAILED DESCRIPTION:
This is a phase I dose-escalation study of oral PCLX-001, conducted in a multicenter, non-randomized, open-label, non-controlled design. The study is comprised of two parts: Part A (single-agent dose escalation) and Part B (single-agent expansion cohorts).

For Part A dose-escalation, patients will be enrolled in cohorts of 3 to 6 patients to each dose level. A new dose level cannot open to accrual until toxicity has been determined in the preceding dose level (i.e. all patients have completed their first cycle of therapy and data for all patients in that dose level have been reviewed at a safety cohort review meeting). Six patients will be treated at the maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D). If required, the MTD cohort may be expanded by an additional 10 patients for further toxicity and response assessment. The MTD cohort expansion may be restricted to B-cell lymphoma or advanced solid tumours to ensure there is proper distribution during dose escalation.

For Part B (single agent expansion cohorts), two expansion cohorts (N=20 each) will be opened to determine the preliminary clinical activity of PCLX-001 at the RP2D:

* Expansion Cohort A: Participants with advanced solid malignancies showing preclinical sensitivity or molecular markers of sensitivity to PCLX-001. This includes breast, nonsmall cell lung (NSCLC), small-cell lung (SCLC), colorectal (CRC), and bladder cancers
* Expansion Cohort B: Participants with relapsed/refractory (R/R) B-cell lymphoma: diffuse large B-cell lymphoma (DLBCL), high grade B-cell lymphoma (HGBL), follicular lymphoma (FL), mantle cell lymphoma (MCL), and Burkitt lymphoma. Transformed large B-cell lymphoma will also be included.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained before any study-specific procedures are performed.
2. Male or female patients aged ≥ 18 years
3. Dose Escalation

   1. Participants with histologically-confirmed advanced solid tumor who have failed at least one prior therapy and/or are not eligible for therapies expected to provide clinical benefit.
   2. Histologically-confirmed B-cell lymphomas that are expected to express CD20 including DLBCL, HGBL, FL (grades 1 to 3b), MCL, and Burkitt lymphoma who have failed at least two prior therapies and/or are not eligible for therapies expected to provide clinical benefit (including autologous stem cell transplantation). Transformed large B-cell lymphoma patients are eligible. FL patients should meet criteria for requiring treatment.

   Dose Expansion Cohort A: Participants with histologically-confirmed advanced breast, NSCLC, SCLC, colorectal, and bladder cancers who have failed at least one prior therapy and/or are not eligible for therapies expected to provide clinical benefit.

   Cohort B: Participants with histologically-confirmed R/R B-cell lymphomas that are expected to express CD20 including DLBCL, HGBL, FL (grades 1-3a), FL (grade 3b), MCL, and Burkitt lymphoma who have failed at least two prior therapies and/or are not eligible for therapies expected to provide clinical benefit. Transformed large B-cell lymphoma patients are eligible. FL patients should meet criteria for requiring treatment.
4. Patients must have evaluable or measurable disease.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
6. Life expectancy of at least 12 weeks
7. Patients must have adequate bone marrow, liver, kidney and cardiac function.
8. Patients must have adequate coagulation.
9. Women of childbearing potential must have a negative pregnancy test.
10. Women of childbearing potential and fertile men must agree to use adequate contraception when sexually active from signing of the informed consent form for the full study until at least 6 months after the last study drug administration.

Exclusion Criteria:

1. Known hypersensitivity to the study drugs or excipients of the preparations or any agent given in association with this study.
2. History of cardiac disease: congestive heart failure New York Heart Association (NYHA) class > II, unstable angina (angina symptoms at rest), new-onset angina (within the past 6 months before study entry), myocardial infarction within the past 6 months before study entry, or uncontrolled cardiac arrhythmias.
3. Uncontrolled arterial hypertension despite optimal medical management.
4. Moderate or severe hepatic impairment.
5. Patients with known human immunodeficiency virus (HIV) infection.
6. Patients who have an active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection requiring treatment.
7. Infections not responding to therapy or active clinically serious infections.
8. Symptomatic metastatic brain or meningeal tumors unless the patient is > 3 months from definitive therapy, has a stable imaging study and is clinically stable. Patients with asymptomatic brain metastases must not be on steroid therapy.
9. Current or past history of central nervous system (CNS) lymphoma.
10. Uncontrolled seizure disorder requiring therapy.
11. History of organ allograft transplantation or autologous stem cell transplantation ≤ 3 months prior to the first dose of study drug. Patients who received prior CAR-T or other T-cell targeting treatment (approved or investigational) ≤ 4 weeks prior to study drug administration.
12. Evidence or history of bleeding disorder within 4 weeks before the first dose of study drug.
13. Serious, non-healing wound, ulcer, or bone fracture.
14. Any malabsorption condition.
15. Breastfeeding. Female patients must not breastfeed during treatment and until 4 months after last study drug administration.
16. Treatment with systemic steroids (prednisone dose ≥10 mg/day or equivalent dose).
17. Acute toxic effects of previous anticancer chemotherapy or immunotherapy that have not yet stabilized or if significant post-treatment toxicities have been observed.
18. Radiotherapy for target lesions during study or within 3 weeks before the first dose of study drug.
19. Major surgery or significant trauma within 4 weeks before the first dose of study drug.
20. Concomitant participation in another clinical study with investigational medicinal product(s).
21. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
22. Use of strong CYP3A4 inhibitors and inducers from 14 days prior to first administration of study drug. Strong CYP3A4 inhibitors and inducers are prohibited during the study and until the active follow up visit.
23. Clinically relevant findings in the ECG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Sangha, Principal Investigator — Cross Cancer Institute
Locations (4):
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - CR Centre Hospitalier de l'Université de Montréal - CHUM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beauchamp E, Yap MC, Iyer A, Perinpanayagam MA, Gamma JM, Vincent KM, Lakshmanan M, Raju A, Tergaonkar V, Tan SY, Lim ST, Dong WF, Postovit LM, Read KD, Gray DW, Wyatt PG, Mackey JR, Berthiaume LG. Targeting N-myristoylation for therapy of B-cell lymphomas. Nat Commun. 2020 Oct 22;11(1):5348. doi: 10.1038/s41467-020-18998-1. PMID 33093447
- [Result] Sangha R, Jamal R, Spratlin J, Kuruvilla J, Sehn LH, Beauchamp E, Weickert M, Berthiaume LG, Mackey JR. A first-in-human phase I trial of daily oral zelenirstat, a N-myristoyltransferase inhibitor, in patients with advanced solid tumors and relapsed/refractory B-cell lymphomas. Invest New Drugs. 2024 Aug;42(4):386-393. doi: 10.1007/s10637-024-01448-w. Epub 2024 Jun 5. PMID 38837078

RESULTS

PARTICIPANT FLOW:
Groups:
- PCLX-001 Intervention 20mg: 20mg daily oral pills for 28 days
- PCLX-001 Intervention 40mg: Drug: PCLX-001 - 40mg
  40mg daily oral pills for 28 days
- PCLX-001 - 70mg: 70mg daily oral pills for 28 days
- PCLX-001 Intervention 100mg: 100mg daily oral pills for 28 days
- PCLX-001 Intervention 140mg: 140mg daily oral pills for 28 days
- PCLX-001 Intervention 210mg: 210mg daily oral pills for 28 days
- PCLX-001 Intervention 280mg: 280mg daily oral pills for 28 days
Period: Overall Study
Arm/Group | PCLX-001 Intervention 20mg | PCLX-001 Intervention 40mg | PCLX-001 - 70mg | PCLX-001 Intervention 100mg | PCLX-001 Intervention 140mg | PCLX-001 Intervention 210mg | PCLX-001 Intervention 280mg
Started | 3 | 3 | 3 | 6 | 3 | 8 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 8 | 3
Not Completed | 0 | 0 | 0 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients were ≥18 years old and had (i) advanced solid tumors with progression after at least one prior therapy and who were not eligible for therapies expected to provide clinical benefit, or (ii) B-cell lymphomas including DLBCL, high grade B-cell lymphoma (HGBL), follicular lymphoma (FL) (grades 1 to 3b), mantle cell lymphoma (MCL), and Burkitt lymphoma who had failed at least two prior therapies.
Groups:
- Total: Total of all reporting groups
Arm/Group | PCLX-001 Intervention 20mg | PCLX-001 Intervention 40mg | PCLX-001 Intervention 70mg | PCLX-001 Intervention 100mg | PCLX-001 Intervention 140mg | PCLX-001 Intervention 210mg | PCLX-001 Intervention 280mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 8 | 3 | 29
Age, Continuous [Median (Full Range); unit: years] | 56 [55 to 86] | 68 [57 to 70] | 66 [61 to 75] | 53 [37 to 69] | 65 [41 to 69] | 56 [37 to 63] | 48 [37 to 63] | 65 [37 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 0 | 5 | 1 | 5 | 2 | 18
  Male | 0 | 1 | 3 | 1 | 2 | 3 | 1 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 2 | 2 | 3 | 6 | 3 | 8 | 3 | 27
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 3 | 3 | 6 | 3 | 8 | 3 | 29
Patients enrolled [Number; unit: participants] | 3 | 3 | 3 | 6 | 3 | 8 | 3 | 29

OUTCOME MEASURES:

1. Primary Outcome: To Determine, During the Dose Escalation Phase, the Recommended Dose of PCLX-001 for the Dose Expansion Phase of the Trial.
Description: The recommended dose will be the dose level below that for the cohort in which maximum tolerated dose (MTD) was reached/exceeded. MTD will have been reached when 2 or more patients in a cohort experience DLT.
Time Frame: Through study completion, an average of ~90 days
Population: Refractory solid tumour and Non-Hodgkins Lymphoma patients for whom no other therapies were available. All evaluable patients were assessed.
Measure: Number; unit: mg
Groups:
- PCLX-001 Intervention: The Dose-Escalation phase will follow a standard 3+3 cohort design. Three patients will be treated at each dose level. If 0/3 patients experience DLT, 3 patients will be treated at the next dose level. Escalation will terminate as soon as two or more patients experience any DLT attributable to study drugs, at a given dose level.
  Oral PCLX-001 will be provided as continuous daily dosing on a 28-day cycle.
  PCLX-001: To ensure maximal safety in this first-in-human trial, the starting dose level was chosen to be 20 mg daily on a 28-day cycle.
Arm/Group | PCLX-001 Intervention
Number analyzed (Participants) | 29
mg | 210

ADVERSE EVENTS:
Time Frame: Through study completion, an average of ~90 days
Description: SAE defined as Grade 3 or higher treatment emergent adverse event.
Arm/Group | PCLX-001 Intervention 20mg | PCLX-001 Intervention 40mg | PCLX-001 Intervention 70mg | PCLX-001 Intervention 100mg | PCLX-001 Intervention 140mg | PCLX-001 Intervention 210mg | PCLX-001 Intervention 280mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 1/6 | 0/3 | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 1/3 | 1/6 | 0/3 | 0/8 | 3/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 0/3 | 0/8 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCLX-001 Intervention 20mg (N=3) | PCLX-001 Intervention 40mg (N=3) | PCLX-001 Intervention 70mg (N=3) | PCLX-001 Intervention 100mg (N=6) | PCLX-001 Intervention 140mg (N=3) | PCLX-001 Intervention 210mg (N=8) | PCLX-001 Intervention 280mg (N=3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroduodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID 19 (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary Disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/95/NCT04836195/Prot_SAP_000.pdf